CLINICAL TRIAL: NCT05972395
Title: Determining if Conditioned Pain Modulation Differs Between Individuals With Localized Versus Widespread Mechanical Pain Hypersensitivity in Chronic Low Back Pain
Brief Title: Conditioned Pain Modulation in Localized vs Widespread Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: LBP01
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Localized CLBP: Chronic low back pain >3 months with localized pressure pain hyperalgesia
  Interventions: Other: Localized vs Widespread Mechanical Pain Hypersensitivity
- Widespread CLBP: Chronic low back pain >3 months with widespread pressure pain hyperalgesia
  Interventions: Other: Localized vs Widespread Mechanical Pain Hypersensitivity

INTERVENTIONS:
Other: Localized vs Widespread Mechanical Pain Hypersensitivity — Based on pressure pain threshold mapping, participants will be classified as having either localized mechanical pain hyperalgesia (hyperalgesia limited to the lumbosacral region) or widespread mechanical pain hyperalgesia (hyperalgesia extending beyond the lumbosacral region).

SUMMARY:
This study aims to compare function of the body's endogenous pain modulation system between people with localized low back pain versus widespread body pain. Endogenous pain modulation refers to the body's natural ability to inhibit one pain stimulus by applying a second pain stimulus. This study will assess pain inhibition by measuring pressure pain thresholds at the low back before and during cold water hand immersion. The researchers hypothesize that those with widespread body pain will have worse functioning of pain inhibition compared to those with localized low back pain only. The results may provide insights into personalized chronic pain management approaches.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is highly prevalent worldwide. Impairments in conditioned pain modulation (CPM) have been documented in CLBP populations. CPM refers to endogenous pain inhibition, where one noxious stimulus inhibits pain from a second noxious stimulus. This relies on descending inhibitory pathways. However, it is unknown whether CPM alterations differ between individuals with localized versus widespread mechanical pain hypersensitivity. The aim of this cross-sectional quantitative sensory testing study is to compare CPM function between localized and widespread CLBP subgroups. A sample of 75 adults with CLBP of at least 3 months duration will be recruited from a chronic pain clinic. Based on pressure pain threshold mapping at the low back and distal sites, participants will be classified as having localized or widespread mechanical hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 years
* Chronic LBP >3 months
* Average LBP intensity ≥4/10

Exclusion Criteria:

* Known LBP pathologies
* Previous lumbar surgery
* Neuropathic LBP
* Comorbid generalized pain conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with chronic nonspecific LBP stratified by localized vs widespread mechanical hyperalgesia
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | Baseline
  Percent change in pressure pain threshold at the lumbar region during cold water hand immersion conditioning stimulus compared to baseline pressure pain threshold at the lumbar region without the conditioning stimulus.

SECONDARY OUTCOMES:
Pressure Pain Thresholds | baseline
  Pressure pain thresholds measured in kg/cm2 using a pressure algometer at the lumbar spine and distal sites including the upper trapezius and thumbnail.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No